CLINICAL TRIAL: NCT05466630
Title: Prospective Evaluation of the Specificity of Serological Tests for Human African Trypanosomiasis in Côte d'Ivoire and Guinea
Brief Title: Prospective Evaluation of the Specificity of Serological Tests for Human African Trypanosomiasis
Acronym: SpeSerTryp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Foundation for Innovative New Diagnostics (Unknown); Programme National de lutte contre la THA, Guinée (Unknown); Université Jean Lorougnon Guédé, Daloa (Unknown); Institut Pasteur, Guinée (Unknown); Institut Pierre Richet, Guinée (Unknown)
Responsible Party: Principal Investigator, Veerle Lejon, Research Director, Institut de Recherche pour le Developpement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SpeSerTryp
Record Dates: First submitted 2022-07-07; First posted 2022-07-20 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Human African Trypanosomiasis; Sleeping Sickness; Trypanosoma Brucei Gambiense; Infection; West African Sleeping Sickness
Keywords: Diagnosis
MeSH Terms: conditions — Trypanosomiasis, African; Infections; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participant (Other): All eligible participants will undergo 5 serological field tests for HAT and a malaria test. Those testing positive in at least 1 serological field test will undergo parasitology to confirm HAT and immunological and molecular laboratory tests
  Interventions: Diagnostic Test: Serological field test for HAT; Diagnostic Test: malaria rapid test; Diagnostic Test: Immunologic laboratory tests; Diagnostic Test: Molecular laboratory tests

INTERVENTIONS:
Diagnostic Test: Serological field test for HAT — Whole blood is tested by lateral flow or agglutination (CATT) for the presence of trypanosome specific antibody. Participants testing positive for at least one of these tests will undergo microscopic examination to detect trypanosomes (lymph, mAECT on blood) and DBS will be prepared for immunological and molecular laboratory testing.
  Other Names: Bioline HAT 2.0 (Abbott, South Korea), HAT Sero-K-SeT (Coris BioConcept, Belgium), HAT 2.0 Sero-K-SeT (Coris BioConcept, Belgium), RDT DCN (USA), CATT/Tb gambiense (ITM Antwerp, Belgium)
Diagnostic Test: malaria rapid test — RDT detecting HRP2 plasmodium antigen.
Diagnostic Test: Immunologic laboratory tests — Laboratory tests detecting trypanosoma brucei gambiense specific (VSG) antibodies in DBS. These tests will only be carried out on participants that are positive in at least on of the rapid serological tests
  Other Names: trypanolysis, ELISA/T.b.gambiense, g-iELISA
Diagnostic Test: Molecular laboratory tests — Laboratory tests detecting Trypanozoon specific nucleic acids. These tests will only be carried out on participants that are positive in at least on of the rapid serological tests
  Other Names: Trypanozoon RT-qPCR multiplex, SNP RT-qPCR, SHERLOCK

SUMMARY:
This study evaluates and compares the diagnostic specificity of 5 serological field tests for screening of the population at risk for human African trypanosomiasis due to Trypanosoma brucei gambiense.

DETAILED DESCRIPTION:
In the last decade, the prevalence of Trypanosoma brucei gambiense (Tbg) human African trypanosomiasis (HAT) has fallen and HAT has been targeted for transmission interruption by 2030. To achieve this goal, disease surveillance remains essential and is based on the identification of cases after screening carried out in the field with a serological test.

The SpeSerTryp study is a prospective evaluation of the specificity of serological field tests for the diagnosis of HAT in Côte d'Ivoire and Guinea. Since the prevalence of HAT is low in these countries, sensitivity will not be assessed.

The main objective is to evaluate and compare the specificity of 5 serological field tests: Bioline HAT 2.0 (Abbott, South Korea), HAT Sero-K-SeT & HAT 2.0 Sero-K-SeT (Coris BioConcept, Belgium ), TDR DCN (USA), and the CATT/T.b. gambiense (Institute of Tropical Medicine Antwerp, Belgium). The secondary objectives are: 1° to assess the specificity of the 5 serological field tests according to malaria status; and 2° to compare the performance of immunological laboratory tests (trypanolysis, ELISA/T.b.gambiense, g-iELISA) and molecular laboratory tests (Trypanozoon RT-qPCR multiplex, SNP RT-qPCR and SHERLOCK) as reference tests to differentiate false positive subjects to serological field tests from subjects who had contact with Tbg. Specificity values will be determined against a composite reference test consisting of the most sensitive HAT parasitological methods. SpeSerTryp is a prospective study that will take place in the endemic health districts of Bonon and Sinfra in Côte d'Ivoire and in the endemic health districts of Forécariah, Dubréka and Boffa in Guinea. In each country, 500 participants will be actively recruited by mobile teams. The inclusion criteria are: Age greater than or equal to 10 years and obtaining signed informed consent. The exclusion criteria are: Severe anemia preventing blood sampling; serious illness preventing the obtaining of informed consent and participation in the study; or history of HAT. After obtaining informed consent, a venous blood sample will be taken (6 mL). This specimen will be used to carry out the 5 serological tests for HAT, the RDT for malaria, and for participants with at least one of the 5 serological tests positive, parasitological confirmation of HAT and molecular and immunological laboratory tests . The duration of participant recruitment is estimated to be around 30 days, while laboratory analyses will take about 6 months. HAT cases identified during the study will be treated in accordance with current national guidelines.

This study will be conducted in accordance with the protocol, the current version of the Declaration of Helsinki, ICH-BPC E6/R2 guidelines, and all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* at least 10 years old
* signed the informed consent form (in case of minor: parent or tutor signs informed consent form and minor signs ascent form)

Exclusion Criteria:

* severe anemia hindering blood sampling
* severe illness hindering obtention of informed consent (eg coma, cognitive deficiency etc)
* history of sleeping sickness

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1095 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Specificity of serological field test for diagnosis of HAT during active screening in Côte d'Ivoire and Guinea | 1 month
  Index tests: Bioline HAT 2.0 (Abbott, South Korea), HAT Sero-K-SeT (Coris BioConcept, Belgium), HAT 2.0 Sero-K-SeT (Coris BioConcept, Belgium), RDT DCN (USA), CATT/Tb gambiense (ITM Antwerp, Belgium). Reference test: parasitological confirmation by combined lymph and blood (mAECT) examination

SECONDARY OUTCOMES:
Specificity of serological field test for diagnosis of HAT during active screening in Côte d'Ivoire and Guinea, in function of malaria status | 1 month
  Index tests: Bioline HAT 2.0 (Abbott, South Korea), HAT Sero-K-SeT (Coris BioConcept, Belgium), HAT 2.0 Sero-K-SeT (Coris BioConcept, Belgium), RDT DCN (USA), CATT/Tb gambiense (ITM Antwerp, Belgium). Reference test: parasitological confirmation by combined lymph and blood (mAECT) examination. The malaria status will be determined using an RDT detecting HRP2
Specificity of immunologic and molecular laboratory tests for diagnosis of HAT in serological suspects | 1 year
  Index tests: trypanolysis, ELISA/T.b.gambiense, g-iELISA, Trypanozoon RT-qPCR multiplex, SNP RT-qPCR, SHERLOCK. Reference test: parasitological confirmation by combined lymph and blood (mAECT) examination.

CONTACTS AND LOCATIONS:
Overall Officials: Martial N'Djetchi Kassi, Principal Investigator — Université Jean Lorougnon Guédé de Daloa; Oumou Camara, Principal Investigator — Programme National de lutte contre de la THA en Guinée
Locations (2):
- Université Jean Lorougnon Guédé de Daloa, Bonon, Côte d’Ivoire
- Programme Nationale de Lutte contre la Trypanosomiase Humaine Africaine, Ministère de Santé, Division Prévention et Lutte contre la Maladie, Dubréka, Guinea

IPD SHARING:
Plan to Share IPD: Yes
As part of the open data policy (FAIR data), the final database of the study will be deposited in the IRD's institutional depository "DataSud" and will be identified by a DOI. Metadata describing the database will be under open access. The database itself, containing personal health data, may be considered "sensitive", and will be under controlled access by a data access committee which will assess specific requests for data use. The partners who generated the data will remain the owners of the data.
Time Frame: Data are estimated to be deposited about 1 year after the start of recruitment. Data will remain available as long as the study is showcased on datasud
Access Criteria: Metadata will be public. Personal health data, may be considered "sensitive", will be under controlled access by a data access committee which will assess specific requests for data use.

REFERENCES:
- [Derived] N'Djetchi MK, Camara O, Koffi M, Camara M, Kaba D, Kabore J, Tall A, Rotureau B, Glover L, Traore MB, Kone M, Coulibaly B, Adingra GP, Soumah A, Gassama M, Camara AD, Compaore CFA, Camara A, Boiro S, Anton EP, Bessell P, Van Reet N, Bucheton B, Jamonneau V, Bart JM, Solano P, Bieler S, Lejon V. Specificity of serological screening tests and reference laboratory tests to diagnose gambiense human African trypanosomiasis: a prospective clinical performance study. Infect Dis Poverty. 2024 Jul 8;13(1):53. doi: 10.1186/s40249-024-01220-5. PMID 38978124